CLINICAL TRIAL: NCT05812833
Title: The Effect of Web-Based Baby Care Education Based on Meleis' Transition Theory on Mother's Self-Confidence and Newborn Health
Brief Title: Web-Based Baby Care Education Meleis' Transition Theory Mother's Self-Confidence Newborn Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Halic University (Other)
Collaborators: Gülçin Bozkurt (Unknown)
Responsible Party: Principal Investigator, Fatma Şule Bilgiç, Lecturer, Halic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: PhD
Record Dates: First submitted 2022-08-03; First posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-03

CONDITIONS: Newborn; Vitality; Theory, Double Bind; Mother-Infant Interaction
Keywords: Meleis Transition Theory; infant health; online education; web page
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Randomized Controlled
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participating in online training and providing active consultancy (Experimental): Online training will be given to mothers, and then the web link will be shared and online counseling will be given every week. Mothers will be followed for 3 months
  Interventions: Behavioral: Education
- Control (No Intervention): Will receive routine maintenance of the institution

INTERVENTIONS:
Behavioral: Education — Pregnant women will be given online baby care training
  Other Names: consultancy
  Arms: Participating in online training and providing active consultancy

SUMMARY:
Web-Based Baby Care Education Meleis' Transition Theory Mother's Self-Confidence Newborn Health

DETAILED DESCRIPTION:
When the mother is not self-confident; They cannot fulfill their motherhood role, have difficulty in establishing a relationship with their baby, and cannot raise their babies in a healthy way. It is easier for mothers who have the necessary knowledge and skills to care for the baby to adapt to this process. The educational support given in the transition to motherhood will affect the mother's self-confidence and readiness for motherhood, thus affecting the baby's health.

The research will be conducted on the online platform between November 2022 and November 2023. The population of the randomized controlled study was Istanbul Haseki Training and Research Hospital Sultan Gazi Haseki Campus, the pregnant women followed in the pregnant outpatient clinic, the sample was n: 45 pregnant women who attended the online training meeting the sample selection criteria, 45 pregnant women informed on the website, and 45 pregnant women in the control group, a total of 135 mothers. will form the candidate. Pregnant women who are willing to participate in the study will be assigned to the groups by simple randomization method. During the research, the CONSORT 2018 statement will be followed. Research data; Data Collection Form will be obtained by Pregnants' Readiness for Newborn Hygienic Care Scale, Karitane Parental Self-Confidence Scale, LACTH (Breastfeeding Success Assessment) Scale and Infant Follow-up Form.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous pregnant
* Single pregnancy
* Expectant mothers with internet access,
* Expectant mothers who can use digital tools (Smartphone or computer)
* Mothers with healthy babies
* Mothers whose babies were born at term (between 37-42 GH)
* Mothers discharged with their baby
* Those whose baby is with the mother
* Expectant mothers who do not attend pregnancy education classes

Exclusion Criteria:

* The mother has communication problems,
* The mother has a chronic illness,
* Having problems with breastfeeding (breast or newborn),

  * The newborn has IUGR or genetic disease,
  * Failure to attend training sessions.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Mother
Enrollment: 135 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Education | 16 weeks
  Web-based online baby care training based on Meleis' Transition Theory to measures mothers' self-confidence
Newborn | 16 weeks
  To evaluate more successful breastfeeding in infants of mothers who received web-based online infant care training based on Meleis' Transition Theory.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Fatih, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Research data collection: 6 months Analysis of data: 3 Months Reporting and publication preparation: 3 Months

REFERENCES:
- [Derived] Bilgic FS, Bozkurt G. The Effect of Online Infant Care Education and Postpartum Counseling Based on Meleis's Transition Theory on Mothers' Self-Esteem and Infant Health: A Randomized Controlled Trial. Nurs Health Sci. 2025 Mar;27(1):e70045. doi: 10.1111/nhs.70045. PMID 39900549